CLINICAL TRIAL: NCT07403032
Title: Study on the Effects and Mechanisms of Modified Ma Xing Shi Gan Decoction in Treating Acute Exacerbations of Chronic Obstructive Pulmonary Disease Based on the "Lung-Large Intestine Mutual Interior-Exterior Relationship"
Brief Title: Study on the Effects and Mechanisms of Modified Ma Xing Shi Gan Decoction in Treating Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cuiling Feng (Other)
Collaborators: Linfen Central Hospital (Unknown); Zhuhai Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Qingyang hospital of traditional Chinese medicine, Gansu Province (Unknown); Traditional Chinese Medicine Hospital of Changji Hui Autonomous Prefecture, Xinjiang (Unknown)
Responsible Party: Sponsor-Investigator, Cuiling Feng, professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025PHB449-001
Record Dates: First submitted 2026-01-12; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: acute exacerbation of chronic obstructive pulmonary disease; modified Ma Xing Shi Gan Decoction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): The patient was given basic Western medical treatment combined with modified Ma Xing Shi Gan Decoction, orally twice a day for 14 days of intervention.
  Interventions: Drug: modified Ma Xing Shi Gan Decoction; Drug: The specific drug comes from "Chinese Expert Consensus on the Diagnosis and Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease (Revised Edition 2023)" and the GOLD guidelines
- control group (Active Comparator): Under the guidance of the "Expert consensus on the acute exacerbation of chronic obstructive pulmonary disease in China (revision in 2023)" and the GOLD guidelines, basic Western medical treatment was given
  Interventions: Drug: The specific drug comes from "Chinese Expert Consensus on the Diagnosis and Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease (Revised Edition 2023)" and the GOLD guidelines

INTERVENTIONS:
Drug: modified Ma Xing Shi Gan Decoction — The patient was given basic Western medical treatment combined with modified Ma Xing Shi Gan Decoction, orally twice a day for 14 days of intervention.
  Arms: test group
Drug: The specific drug comes from "Chinese Expert Consensus on the Diagnosis and Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease (Revised Edition 2023)" and the GOLD guidelines — Under the guidance of the "Expert consensus on the acute exacerbation of chronic obstructive pulmonary disease in China (revision in 2023)" and the GOLD guidelines, basic Western medical treatment was given. The main types include third-generation cephalosporins, expectorants, short-acting anticholinergic drugs, and short-acting β2 receptor agonists, etc.

SUMMARY:
This study adopted a multi-center, randomized, controlled trial design. Patients with acute exacerbation of chronic obstructive pulmonary disease who met the inclusion criteria were randomly assigned to the experimental group and the control group. Both groups were treated under the guidance of the "Expert consensus on the acute exacerbation of chronic obstructive pulmonary disease in China (revision in 2023)" and the GOLD guidelines. The experimental group was treated with modified Maxing Shigan Decoction. The modified Ma Xing Shi Gan Decoction was administered twice a day for 14 days. Taking the length of hospital stay (days) of the patients as the primary efficacy indicator, and the TCM syndrome score, dyspnea score (mMRC), 6-minute walk test and mechanical ventilation demand rate as the secondary efficacy indicators, the clinical efficacy of modified Maxing Shigan Decoction in the treatment of acute exacerbation of chronic obstructive pulmonary disease was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting diagnostic criteria for COPD exacerbation, as defined by "Expert consensus on the acute exacerbation of chronic obstructive pulmonary disease in China (revision in 2023)" ;
2. Patients meeting the diagnostic criteria for phlegm-heat stagnation in the lungs syndrome within COPD, as referenced in the "Clinical Diagnosis and Treatment Terminology of Traditional Chinese Medicine: Syndromes" and the 2020 International Guidelines for Clinical Practice of Traditional Chinese Medicine;
3. Age > 18 years;
4. Hospitalized patients;
5. Voluntarily consent to treatment and sign an informed consent form.

Exclusion Criteria:

1. History of allergy to the study drug;
2. History of active liver disease;
3. Patients undergoing dialysis or with known moderate to severe renal impairment;
4. Suspected or confirmed active systemic infection;
5. Patients with host immune dysfunction, host immunodeficiency, or host immune reconstitution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay (days) | collected at baseline, 7 days, and 14 days post-treatment.
  Number of days the patient remains hospitalized during the study period.

SECONDARY OUTCOMES:
Traditional Chinese Medicine symptom score | collected at baseline, 7 days, and 14 days post-treatment
  The Traditional Chinese Medicine Syndrome Rating Scale is divided into four severity levels: absent, mild, moderate, and severe. Primary symptoms include cough, sputum volume, sputum characteristics, chest fullness and oppression, and dyspnea. Scores range from 0 (least severe) to 6 (most severe). Secondary symptoms include fever, restlessness, thirst with desire to drink, and urinary and bowel status. Scores range from 0 to 3 based on severity. The sum of these scores constitutes the total score. A higher total score indicates greater severity.
Dyspnea assessment | collected at baseline, 7 days, and 14 days post-treatment.
  mMRC questionnaire
Mechanical Ventilation Requirement Rate | collected at baseline, 7 days, and 14 days post-treatment.
  Data is collected in real-time via the hospital's Electronic Medical Record (EMR) system and the ICU ventilator recording system to calculate Total Mechanical Ventilation Time (TMVT). This is further analyzed to distinguish Invasive Mechanical Ventilation Time (IMVT) and Non-Invasive Mechanical Ventilation Time (NIMVT).
6-Minute Walk Test Distance | Measured at baseline, 7 days, and 14 days.
Complete blood count (CBC) | Collected at baseline, 7 days, and 14 days.
C-reactive protein (CRP) | collected at baseline, 7 days, and 14 days post-treatment.

IPD SHARING:
Plan to Share IPD: Undecided
have not decided